CLINICAL TRIAL: NCT03139032
Title: A Phase 2a, Proof of Concept, Open-label Study Evaluating the Efficacy and Safety of Etrasimod (APD334) in Inflammatory Bowel Disease Patients With Active Skin Extra-intestinal Manifestations
Brief Title: Efficacy and Safety of Etrasimod (APD334) in Inflammatory Bowel Disease Patients With Active Skin Extra-intestinal Manifestations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate the study
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APD334-006
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Inflammatory Bowel Diseases; Skin Extra-intestinal Manifestations
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — etrasimod

STUDY DESIGN:
Intervention Model Description: Proof of concept, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APD334 (Experimental): APD334 active treatment for 12 weeks.
  Interventions: Drug: APD334

INTERVENTIONS:
Drug: APD334 — APD334 active treatment for 12 weeks.
  Other Names: Etrasimod

SUMMARY:
The purpose of this phase 2a, proof of concept, open-label clinical study is to evaluate the efficacy and safety of etrasimod (APD334) in inflammatory bowel disease patients with active skin extra-intestinal manifestations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (18-80 years).
2. Able to provide a signed informed consent prior to any study related procedure being conducted.
3. Considered to be in stable health in the opinion of the investigator as determined by:

   1. A pre-study physical examination with no clinically significant abnormalities unrelated to IBD.
   2. Vital signs at screening: pulse rate ≥ 55 bpm, systolic blood pressure ≥ 90, and diastolic blood pressure ≥ 55 mmHg.
   3. Liver function tests (ALT/AST, bilirubin and alkaline phosphatase) < 2x the upper limit of normal.
   4. All other pre-study clinical laboratory findings within normal range, or if outside of the normal range are not deemed clinically significant in the opinion of the investigator.
   5. 12-lead electrocardiogram showing no clinically significant abnormalities in the opinion of the investigator (for confirmation please refer to exclusion criterion # 22).
   6. A chest x- ray showing no evidence of active pulmonary disease (a chest x-ray taken within the previous 12 months from the screening visit may also be used).
   7. Ophthalmology evaluation (by an ophthalmologist) without evidence of macular edema, supported with optical coherence tomography where available (dependent on site capability) no later than 3 months prior to screening.
4. Patients receiving stable treatment for IBD and EIM.
5. Diagnosis of active psoriasis, erythema nodosum or pyoderma gangrenosum by Investigator assessments. After the enrollment of 10 patients with active EIM, patients with active psoriasis due to anti TNF-alpha therapy can also be included.
6. Diagnosis of ulcerative colitis or Crohn's disease established prior to screening by clinical and endoscopic evidence.
7. Eligible male and female patients must agree not to participate in a conception process (i.e. active attempt to let female partner to become pregnant or to impregnate, sperm donation, oocyte donation, in vitro fertilization) for at least 30 days after the last dose of study drug.

Non-sterile patients who are sexually active must take adequate contraception measures.

Exclusion Criteria:

1. Evidence of abdominal abscess or toxic megacolon at the screening visit.
2. Patients with history of extensive colitis or pancolitis (duration > 8 years) or left-sided colitis (duration > 12 years) must have documented evidence that a surveillance colonoscopy was performed within 12 months of the initial screening visit (if not, the patient should undergo a colonoscopy in lieu of a flexible proctosigmoidoscopy during screening).
3. Previous extensive colonic resection (subtotal or total colectomy).
4. Current evidence of adenomatous colonic polyps that have not been removed.
5. Current evidence of colonic mucosal dysplasia.
6. Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine or stoma.
7. Clinical significant infection as judged by the investigator in the previous 6 weeks before enrollment.
8. Evidence of or treatment for C. difficile infection within 60 days, or other intestinal pathogen within 30 days, prior to randomization.
9. Exposure to natalizumab or rituximab within 5 half-lives prior to randomization.
10. Treatment of underlying disease within 30 days prior to randomization (5-ASA, corticosteroids, TNF-alpha inhibitors, probiotics, antidiarrheals, azathioprine and 6-mercaptopurine may be allowed under certain conditions).
11. Receipt of any investigational agent within 30 days or 5 half-lives (whichever is longer) prior to randomization.
12. Currently require or are anticipated to require surgical intervention for IBD during the study.
13. Abnormal (< 80% of predicted values) forced expiratory volume (FEV1) or forced vital capacity (FVC).
14. Infection with hepatitis C virus anytime in the past; confirmed active infection with hepatitis B virus at screening.
15. Active or latent tuberculosis (TB), regardless of treatment history, as evidenced by any of the following:

    1. History of TB
    2. A positive diagnostic TB test within one month of randomization
    3. Chest X-ray within 12 months of randomization in which active or latent TB cannot be excluded.
16. Any known history of congenital or acquired immunodeficiency.
17. Clinically significant extra-intestinal infection (e.g., pneumonia, pyelonephritis) within 30 days prior to randomization.
18. Recent history (within 6 months of screening visit) of cardio- or cerebrovascular disease, acute coronary syndrome, myocardial infarction, unstable angina, cerebro-vascular accident, including transient ischemic attack.
19. Any surgical procedure requiring general anesthesia within 30 days prior to randomization or plans to undergo major surgery during the study period.
20. History of retinal macular edema.
21. History of or signs and symptoms of progressive multifocal leukoencephalopathy (PML) as assessed by the PML checklist.
22. History or presence of cardiac arrhythmia, conduction system disease, or use of Class Ia or Class III anti arrhythmic agents, or baseline QTc ≥ 500 msec.
23. Infection requiring hospitalization or intravenous antimicrobial therapy, or opportunistic infection within 4 weeks of screening.
24. History of more than one episode of herpes zoster or any episode of disseminated zoster.
25. Without documented positive varicella zoster virus (VZV) IgG antibody status or who have completed VZV vaccination within 30 days prior to randomization.
26. Receipt of live vaccine within 4 weeks prior to screening.
27. History of lymphoproliferative disorder, lymphoma, leukemia, myeloproliferative disorder, or multiple myeloma.
28. History of malignancy except for adequately treated basal cell skin cancer.
29. History of severe allergic or anaphylactic reactions requiring medical attention.
30. Current or recent history (within one year prior to randomization) of alcohol dependence or illicit drug use.
31. History of clinically significant leukopenia or lymphopenia at screening.
32. Active psychiatric problems that, in the investigator's opinion, may interfere with compliance with the study procedures.
33. History of any clinically significant medical condition that, in the investigator's opinion, would preclude participation in the study.
34. Use of moderate to strong inhibitors of CYP2C9.
35. History of severe renal or hepatic impairment.
36. Inability to attend all the study visits or comply with study procedures.
37. Prior exposure to etrasimod (APD334).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Arena 2001, Leuven, Belgium
- Arena 1001, Hamburg, Germany
- Arena 3001, Belgrade, Serbia

RESULTS

PARTICIPANT FLOW:
Groups:
- Etrasimod: Participants received active treatment for 12 weeks.
Period: Overall Study
Arm/Group | Etrasimod
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Etrasimod
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants]
  Between 18 to 80 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Reporting demographic results for this study in which a single participant was enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
  Male | NA — Reporting demographic results for this study in which a single participant was enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | NA — The demographics of the study doesn't support the reporting of results for a single participant without running a risk of participant re-identification. In order to protect the participant's privacy, results for this study cannot be reported.
  Not Hispanic or Latino | NA — The demographics of the study doesn't support the reporting of results for a single participant without running a risk of participant re-identification. In order to protect the participant's privacy, results for this study cannot be reported.
  Unknown or Not Reported | NA — The demographics of the study doesn't support the reporting of results for a single participant without running a risk of participant re-identification. In order to protect the participant's privacy, results for this study cannot be reported.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — The demographics of the study doesn't support the reporting of results for a single participant without running a risk of participant re-identification. In order to protect the participant's privacy, results for this study cannot be reported.
  Asian | NA — The demographics of the study doesn't support the reporting of results for a single participant without running a risk of participant re-identification. In order to protect the participant's privacy, results for this study cannot be reported.
  Native Hawaiian or Other Pacific Islander | NA — The demographics of the study doesn't support the reporting of results for a single participant without running a risk of participant re-identification. In order to protect the participant's privacy, results for this study cannot be reported.
  Black or African American | NA — The demographics of the study doesn't support the reporting of results for a single participant without running a risk of participant re-identification. In order to protect the participant's privacy, results for this study cannot be reported.
  White | NA — The demographics of the study doesn't support the reporting of results for a single participant without running a risk of participant re-identification. In order to protect the participant's privacy, results for this study cannot be reported.
  More than one race | NA — The demographics of the study doesn't support the reporting of results for a single participant without running a risk of participant re-identification. In order to protect the participant's privacy, results for this study cannot be reported.
  Unknown or Not Reported | NA — The demographics of the study doesn't support the reporting of results for a single participant without running a risk of participant re-identification. In order to protect the participant's privacy, results for this study cannot be reported.

OUTCOME MEASURES:

1. Primary Outcome: Exploratory Endpoint - Change From Baseline in Endoscopic Improvement/Histologic Healing Using Endoscopy or Flexible Proctosigmoidoscopy
Description: Only if there are signs of inflammation at screening another evaluation was planned to be performed at week 12.
Time Frame: Weeks 12
Population: Efficacy analyses were not conducted due to low enrollment (N=1). In order to protect participant's privacy, the results from a single participant cannot be reported.
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

2. Primary Outcome: Exploratory Endpoint - Change From Baseline in Level of Fecal Calprotectin
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

3. Primary Outcome: Exploratory Endpoint - Change From Baseline in Physician Global Assessments for Active Skin Extra-intestinal Manifestations (EIM) (PG, EN and Psoriasis)
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

4. Primary Outcome: Exploratory Endpoint - Change From Baseline in Patient Global Assessments for Active Skin EIM
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

5. Primary Outcome: Exploratory Endpoint - Change From Baseline in the Dermatology Life Quality Index Score
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

6. Primary Outcome: Exploratory Endpoint - Change From Baseline in Inflammatory Bowel Disease Questionnaire Score
Time Frame: Weeks 2, 4, 8, and 12
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

7. Primary Outcome: Exploratory Endpoint - Change From Baseline in C-reactive Protein
Time Frame: Weeks 1, 2, 4, 8, 12 and the 2-week follow-up visit
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

8. Primary Outcome: Exploratory Endpoint - Change From Baseline in Leucocyte Characterization
Time Frame: Weeks 8 and 12
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

9. Primary Outcome: Exploratory Endpoint - Change From Baseline in Stool Frequency at Ulcerative Colitis Endpoint
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

10. Primary Outcome: Exploratory Endpoint - Change From Baseline in Rectal Bleeding at Ulcerative Colitis Endpoint
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

11. Primary Outcome: Exploratory Endpoint - Change From Baseline in Physicians Global Assessments at Ulcerative Colitis Endpoint
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

12. Primary Outcome: Exploratory Endpoint - Change From Baseline in Lymphocyte Counts
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: as for outcome 1
Groups:
- Etrasimod: Participants received one active treatment for 12 weeks.
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

13. Primary Outcome: Exploratory Endpoint - Change From Baseline in Disease Activity Score at Crohn's Disease Endpoint
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

14. Primary Outcome: Exploratory Endpoint - Change From Baseline in Psoriasis Area and Severity Index at Psoriasis Endpoint
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

15. Primary Outcome: Exploratory Endpoint - Changes in Degree of Immune Cell Infiltration as Assessed From Skin Punch Biopsies (From Healthy Skin and From Target Lesion)
Time Frame: Weeks -1, 8, and 12.
Population: Efficacy analyses were not conducted due to low enrollment (N=1). To protect participant's privacy, the results from a single participant cannot be reported.
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

16. Primary Outcome: Exploratory Endpoint -Changes in Levels of Cytokine Expression as Assessed From Skin Punch Biopsies (From Healthy Skin and From Target Lesion)
Time Frame: Weeks -1, 8 and 12.
Population: as for outcome 1
Arm/Group | Etrasimod
Number analyzed (Participants) | 0

17. Other Pre Specified Outcome: Safety Measured by Number of Participants With Adverse Events and Serious Adverse Events
Description: Planned safety evaluations included clinical laboratory tests (chemistry, hematology, and urinalysis), vital signs (blood pressure, pulse, respiratory rate, and oral temperature), physical examination (assessment of general appearance, skin, head [eyes, ears, nose and throat], neck, thyroid, lungs, heart, abdomen, back, lymph nodes, and extremities, and body weight), 12-lead electrocardiograms, adverse event reporting, concomitant medication, and lymphocyte counts.
Time Frame: From date of first dose of study treatment to the safety follow-up visit, approximately 14 weeks
Population: There were no analysis populations in the single participant study. Safety results for the single participant are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Etrasimod
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment until the follow-up safety visit, approximately 14 weeks.
Arm/Group | Etrasimod
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Due to limited enrollment (N=1), this clinical trial was terminated by the Sponsor and no efficacy analyses were conducted. To protect the single participant's privacy, demography and efficacy data are not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT03139032/Prot_SAP_000.pdf